CLINICAL TRIAL: NCT00625183
Title: A Phase II Study of Capecitabine, Oxaliplatin and Selenomethionine and Radiation Therapy in Patients With Stage II and III Rectal Adenocarcinoma
Brief Title: Capecitabine, Oxaliplatin, Selenomethionine, and Radiation Therapy in Treating Patients Undergoing Surgery For Newly Diagnosed Stage II or III Rectal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to poor/low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 113607; RPCI-I-113607
Record Dates: First submitted 2008-02-26; First posted 2008-02-28 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Selenomethionine; Capecitabine; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

ARMS (1):
- Capecitabine, Oxaliplatin, Selenomethionine, Radiation Therapy (Experimental): Oxaliplatin: 50 mg/m2 weekly x 5 Capecitabine 725 mg/m2BID on days of RT Selenomethionine: 4000mcg/m2 PO BID X 7 days prior to RT, then 4000mcg/m2 PO QD from first to last day of RT, including weekends
  Interventions: Dietary Supplement: selenomethionine; Drug: capecitabine; Drug: oxaliplatin; Other: laboratory biomarker analysis; Other: pharmacological study; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: selenomethionine
Drug: capecitabine
Drug: oxaliplatin
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Selenomethionine may slow the growth of tumor cells. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together With selenomethionine and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well selenomethionine works when given together with capecitabine, oxaliplatin, and radiation therapy in treating patients undergoing surgery for newly diagnosed stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete pathological response rate of the combination of capecitabine, oxaliplatin, selenomethionine, and radiotherapy in patients with stage II or III rectal adenocarcinoma.
* To determine the T-downstaging rate with this regimen in patients with stage II or III rectal adenocarcinoma.

Secondary

* To determine the safety of this regimen by assessing toxicity and dose intensity of the various components of this regimen.
* To determine the rate of local relapse.
* To determine the rate of distant relapse.

OUTLINE: Patients receive neoadjuvant therapy comprising oral selenomethionine twice daily for 1 week prior to radiotherapy and then once daily for 6 weeks. Patients also receive oxaliplatin IV over 2 hours on days 1-7 and oral capecitabine twice daily on days 1-5 for 6 weeks and undergo radiotherapy 5 days a week for 6 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

Within 4-8 weeks after completion of neoadjuvant therapy, patients undergo curative-intent surgery. Beginning 4-8 weeks after surgery, patients may receive up to 9 courses of standard adjuvant combination chemotherapy (FOLFOX).

Blood samples are collected at baseline and weekly during treatment and analyzed by absorption spectrophotometry for selenium measurement of drug concentration. Pharmacokinetic studies are also performed.

After completion of study treatment, patients are followed for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed rectal adenocarcinoma that is involving the distal 12 cm of the rectum (above the anal verge)

  * Staged within 8 weeks prior to initiation of study by endoscopic ultrasound OR MRI or CT scan if endorectal ultrasound is non-conclusive or non-tolerable
  * T3-T4 tumor or evidence of lymph node involvement defined by the presence of at least 1 enlarged peri-rectal lymph node
* No evidence of distant or known metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 1 year
* Leukocytes ≥ 3,000/µL
* Absolute neutrophil count ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Total bilirubin ≤ upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* Creatinine ≤ ULN OR creatinine clearance ≥ 60 mL/min
* Able to receive oral medication
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent or previous malignancies unless disease free for > 5 years (excluding nonmelanoma skin cancer)
* No neuropathy ≥ grade 2
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to oxaliplatin, capecitabine, or selenomethionine
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the pelvis
* No prior chemotherapy
* No other concurrent investigational or anticancer agents or therapies
* No concurrent vitamin B6 supplementation (except as part of a standard, multivitamin supplement)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther: Oxaliplatin: 50 mg/m2 weekly x 5 Capecitabine 725 mg/m2BID on days of RT Selenomethionine: 4000mcg/m2 PO BID X 7 days prior to RT, then 4000mcg/m2 PO QD from first to last day of RT, including weekends
Period: Overall Study
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther
Started | 5
Completed | 4
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.48 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathological Response Rate
Time Frame: After completion of capecitabine, oxaliplatin, selenomethionine, and radiation, and before surgery. Assessed endoscopically.
Population: Due to the study's early termination, as a result of low accrual, target accrual was not reached and no data was not collected for this assessment.
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine, Radiation Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Rate of T-downstaging With Capecitabine, Oxaliplatin, Selenomethionine, and Radiotherapy
Time Frame: as for outcome 1
Population: Due to the study's early termination, as a result of low accrual, target accrual was not reached and no data was collected for this assessment.
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine, Radiation Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Safety and Tolerability as Assessed by NCI CTCAE Version 3.0
Description: Number of participants with any adverse event as assessed by NCI CTCAE version 3.0.
Time Frame: Adverse events were queried for and collected every cycle for the duration of treatment.
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine, Radiation Therapy
Number analyzed (Participants) | 5
Participants | 5

4. Secondary Outcome: Dose Intensity
Time Frame: During treatment with capecitabine, oxaliplatin, selenomethionine.
Population: as for outcome 2
Groups:
- Capecitabine, Oxaliplatin, Selenomethionine,Radiation Therapy: Oxaliplatin: 50 mg/m2 weekly x 5 Capecitabine 725 mg/m2BID on days of RT Selenomethionine: 4000mcg/m2 PO BID X 7 days prior to RT, then 4000mcg/m2 PO QD from first to last day of RT, including weekends
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine,Radiation Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Local Relapse Rate
Time Frame: For up to 5 years following surgery.
Population: as for outcome 2
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther
Number analyzed (Participants) | 0

6. Secondary Outcome: Distant Relapse Rate
Time Frame: For up to 5 years following surgery.
Population: as for outcome 1
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine,Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther (N=5)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine, Oxaliplatin, Selenomethionine and Radiation Ther (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (6)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 5 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 4 (6)
Hypersensitivity (Immune system disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7)
Dysgeusia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination, as a result of low accrual, target accrual was not reached and no statistical inference of the primary and secondary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes